CLINICAL TRIAL: NCT03718065
Title: Impact of Lofexidine on Stress, Craving and Opioid Use
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Pro00081381; 2U54DA016511-16 (NIH)
Record Dates: First submitted 2018-10-23; First posted 2018-10-24 (Actual); Results first posted 2025-02-07 (Actual); Last update posted 2025-02-07 (Actual); Status verified 2025-02

CONDITIONS: Opioid-use Disorder; Opiate Dependence
MeSH Terms: conditions — Opioid-Related Disorders | interventions — lofexidine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Lofexidine Men (Experimental): Men will receive lofexidine (Lucemyra) for 5 weeks. Titration schedule is as follows: 0.36 mg on the first two evenings, 0.36 mg in the morning and evening on days 3 and 4; 0.36 mg in the morning, afternoon, and at bedtime on days 5 and 6; 0.36 mg in the morning and afternoon and 0.72 mg at bedtime on days 7 and 8; 0.36 mg in the morning and 0.72 mg in the afternoon and at bedtime on days 9 and 10, and 0.72 mg in the morning, afternoon and at bedtime on Day 11 and throughout the rest of the study.
  Interventions: Drug: Lofexidine
- Lofexidine Women (Experimental): Women will receive lofexidine (Lucemyra) for 5 weeks. Titration schedule is as follows: 0.36 mg on the first two evenings, 0.36 mg in the morning and evening on days 3 and 4; 0.36 mg in the morning, afternoon, and at bedtime on days 5 and 6; 0.36 mg in the morning and afternoon and 0.72 mg at bedtime on days 7 and 8; 0.36 mg in the morning and 0.72 mg in the afternoon and at bedtime on days 9 and 10, and 0.72 mg in the morning, afternoon and at bedtime on Day 11 and throughout the rest of the study.
  Interventions: Drug: Lofexidine
- Placebo Men (Placebo Comparator): Men will receive matching placebo for five weeks.
  Interventions: Drug: Placebo
- Placebo Women (Placebo Comparator): Women will receive matching placebo for five weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Lofexidine — Lofexidine, sold under the brand name Lucemyra among others, is a medication historically used to treat high blood pressure, but more commonly used to help with the physical symptoms of opioid withdrawal. It is taken by mouth. It is an α2A adrenergic receptor agonist.
  Other Names: Lucemyra
  Arms: Lofexidine Men; Lofexidine Women
Drug: Placebo — Placebo comparator.
  Arms: Placebo Men; Placebo Women

SUMMARY:
Individuals with opioid use disorder who are stabilized on buprenorphine or methadone will be randomly assigned to receive placebo or lofexidine for 5 weeks. At the end of five weeks, they will complete a human laboratory stress task and scripted opioid imagery task. Throughout the study a CREMA app (Cue Reactivity Ecological Momentary Assessment) will be used to monitor stress, craving and use in the natural environment.

DETAILED DESCRIPTION:
Participants will complete a screening visit to determine study eligibility. During the first week, participants will be asked to abstain from opioid use other than buprenorphine. Participants will come to the clinic 2 times that week for urine drug testing. If all 2 tests are negative, participants will be randomly assigned to take either lofexidine or placebo (inactive medication) two to three times a day for 5 weeks. During this time, participants will upload videos of themselves taking their medication. They will come to the clinic 3 times a week for urine drug screens and to have their vital signs measured. They will also participate in "CREMA" sessions (Cue Reactivity Ecologic Momentary Assessment) 3 times a day. These sessions include looking at stressful and neutral pictures and rating stress and craving. At the end of five weeks, participants will return to the clinic and participate in a stress task and a scripted opioid imagery task the following day. For the next five days, participants will taper their medication dose. During this time they will continue to come to clinic to have their vital signs measured and complete a follow-up visit.

ELIGIBILITY:
Inclusion Criteria

1. Able to provide informed consent and function at an intellectual level sufficient to allow accurate completion of all assessment instruments.
2. Meet DSM-5 criteria for opioid use disorder (within the past three months). While individuals may also meet criteria for mild use disorders of other substances, they must identify opioids as their primary substance of abuse and must not meet criteria for any other moderate or severe substance use disorder (except tobacco, caffeine, or marijuana) within the last 60 days.
3. On a stable dose of daily buprenorphine or methadone for at least 2 weeks.
4. Age 18-65.
5. Women of childbearing potential must agree to use an effective means of birth control.
6. Consent to remain abstinent from opioids during the 1-week baseline assessment period.
7. Must consent to random assignment.

Exclusion Criteria

1. Women who are pregnant, nursing or of childbearing potential and not practicing an effective means of birth control.
2. Evidence or history of major medical illnesses, including liver diseases, abnormal vaginal bleeding, suspected or known malignancy, thrombophlebitis, deep vein thrombosis, pulmonary embolus, clotting or bleeding disorders, heart disease, insulin-dependent diabetes, history of stroke or other medical conditions that the investigator deems as contraindicated for the individual to be in the study.
3. History of or current psychotic disorder or bipolar I affective disorder.
4. Current suicidal or homicidal ideation/risk.
5. Taking medications known to act on adrenergic systems (B-blockers; alpha agonists or antagonists)
6. Hypotensive individuals with a sitting blood pressure of < 90/50
7. QTc interval of >440 in males and > 460 in females as the combination of lofexidine plus buprenorphine may increase the QTc interval.
8. Known allergy to lofexidine
9. Unable to comply with study procedures or pose threat to study staff.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 112 (Actual)
Dates: Start 2019-06-26 (Actual); Primary Completion 2024-01-30 (Actual); Study Completion 2024-01-30 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Medical University of South Carolina, Charleston, South Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Guille C, King C, Ramakrishnan V, Baker N, Cortese B, Nunn L, Rogers T, McRae-Clark A, Brady K. The impact of lofexidine on stress-related opioid craving and relapse: Design and methodology of a randomized clinical trial. Contemp Clin Trials. 2021 Dec;111:106616. doi: 10.1016/j.cct.2021.106616. Epub 2021 Nov 2. PMID 34737091

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Lofexidine Men | Lofexidine Women | Placebo Men | Placebo Women
Started | 35 | 24 | 24 | 29
Completed | 30 | 18 | 23 | 25
Not Completed | 5 | 6 | 1 | 4

BASELINE CHARACTERISTICS:
Population: The baseline population is all participants who were randomized and began taking medication. Due to participant attrition, the N's for outcome measures are slightly lower.
Groups:
- Total: Total of all reporting groups
Arm/Group | Lofexidine Men | Lofexidine Women | Placebo Men | Placebo Women | Total
Number analyzed (Participants) | 35 | 24 | 24 | 29 | 112
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 35 | 24 | 24 | 29 | 112
  >=65 years | 0 | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 38 (9.17) | 35.79 (7.34) | 40.71 (9.70) | 35.34 (7.51) | 37.42 (8.65)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 24 | 0 | 29 | 53
  Male | 35 | 0 | 24 | 0 | 59
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 1 | 1 | 4 | 1 | 7
  White | 34 | 23 | 20 | 28 | 105
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 35 | 24 | 24 | 29 | 112

OUTCOME MEASURES:

1. Primary Outcome: Drug Cue+ Stressor Induced Craving
Description: Participants will rate craving on a 0 to 7 Likert scale with 0 indicate "Strongly disagree" that they crave and 7 indicating "strongly agree" that they crave so that higher scores indicate more craving.
Time Frame: Pre- Cue and 0, 5, 30 and 60 minutes Post-Cue 5 weeks Post- Baseline; Pre-TSST and 0, 5, 30 and 60 minutes Post-TSST 5 weeks Post-Baseline
Population: Participants with available data on the Trier Social Stress Task (TSST) or Scripted Imagery Cue (Cue). TSST and Cue Tasks were counterbalanced.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Lofexidine Men | Lofexidine Women | Placebo Men | Placebo Women
Number analyzed (Participants) | 27 | 19 | 22 | 23
units on a scale
  Pre-Cue | 1.52 (1.56) | 1 (0) | 1.72 (1.69) | 1.96 (1.61)
  Cue + 0 Minutes | 2.33 (2.06) | 3.58 (2.97) | 2.05 (2.10) | 3.56 (2.54)
  Cue + 5 Minutes | 2 (1.75) | 2.74 (3.02) | 1.86 (1.73) | 2.83 (2.35)
  Cue + 30 Minutes | 1.56 (1.48) | 1.68 (1.67) | 1.77 (1.57) | 2.09 (2.13)
  Cue + 60 Minutes | 1.48 (1.37) | 1.32 (0.95) | 1.86 (1.73) | 1.87 (2.07)
  Pre-TSST | 1.39 (0.69) | 1.11 (0.32) | 1.68 (1.58) | 2.19 (2.02)
  TSST + 0 Minutes | 1.64 (1.31) | 2.72 (2.16) | 2.27 (2.33) | 2.95 (2.78)
  TSST + 5 Minutes | 1.64 (1.45) | 1.89 (1.23) | 2 (1.8) | 2.52 (2.36)
  TSST + 30 Minutes | 1.36 (0.95) | 1.18 (0.39) | 1.82 (1.59) | 2.33 (2.27)
  TSST + 60 Minutes | 1.57 (1.83) | 1.24 (0.44) | 1.77 (1.69) | 2.24 (2.14)

2. Primary Outcome: Drug Cue+ Stressor Induced Stress Response
Description: Participants will rate stress on a 0 to 4 Likert scale with 0 indicate "not at all" and 4 indicating "extremely" so that higher scores indicate a more robust stress response.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Lofexidine Men | Lofexidine Women | Placebo Men | Placebo Women
Number analyzed (Participants) | 27 | 19 | 22 | 21
units on a scale
  Pre-Cue | 2.81 (2.63) | 2.74 (1.66) | 2.77 (2.22) | 2.65 (2.33)
  Cue + 0 Minutes | 3.70 (2.85) | 5.37 (2.81) | 3.23 (2.6) | 3.61 (2.31)
  Cue + 5 Minutes | 2.78 (2.53) | 4.16 (3.08) | 2.68 (2.06) | 3.09 (2)
  Cue + 30 Minutes | 2.56 (2.5) | 2.74 (2.05) | 2.59 (2.21) | 2.30 (1.74)
  Cue + 60 Minutes | 2.63 (2.64) | 2.38 (1.45) | 2.64 (2.34) | 2.61 (2.19)
  Pre-TSST | 2.57 (2.15) | 2.61 (1.75) | 3 (2.18) | 2.57 (1.89)
  TSST + 0 Minutes | 4.89 (3.41) | 5.78 (2.90) | 3.86 (2.55) | 4.95 (3.12)
  TSST + 5 Minutes | 3.54 (3.05) | 3.61 (1.97) | 2.82 (2.26) | 3.10 (1.87)
  TSST + 30 Minutes | 3.04 (3.01) | 2.47 (1.33) | 2.82 (2.02) | 2.76 (1.95)
  TSST + 60 Minutes | 2.89 (2.71) | 2.41 (1.46) | 2 (1.95) | 2.52 (1.47)

ADVERSE EVENTS:
Time Frame: Baseline to end of study taper- 6 weeks.
Arm/Group | Lofexidine Men | Lofexidine Women | Placebo Men | Placebo Women
All-Cause Mortality (participants affected / at risk) | 0/35 | 0/24 | 0/24 | 0/29
Serious Adverse Events (participants affected / at risk) | 0/35 | 0/24 | 0/24 | 0/29
Other Adverse Events (participants affected / at risk) | 28/35 | 17/24 | 10/24 | 13/29
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lofexidine Men (N=35) | Lofexidine Women (N=24) | Placebo Men (N=24) | Placebo Women (N=29)
Dry Mouth (Endocrine disorders) | 18 (21) | 12 (13) | 4 (4) | 5 (5)
Tiredness/Drowsiness (Nervous system disorders) | 15 (17) | 8 (10) | 3 (3) | 4 (6)
Dizziness (Nervous system disorders) | 7 (7) | 2 (2) | 2 (2) | 1 (1)
Headache (Nervous system disorders) | 6 (6) | 5 (5) | 3 (3) | 6 (7)
Fatigue (Nervous system disorders) | 5 (5) | 6 (7) | 0 (0) | 1 (1)
Nausea (Nervous system disorders) | 3 (3) | 0 (0) | 0 (0) | 2 (2)
Lightheadedness (Nervous system disorders) | 3 (3) | 2 (2) | 0 (0) | 1 (1)
Sweating (Nervous system disorders) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 2 (2) | 0 (0) | 1 (1) | 2 (2)
Anxiety (Nervous system disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Grogginess (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2023-07-25): https://cdn.clinicaltrials.gov/large-docs/65/NCT03718065/Prot_SAP_ICF_000.pdf